CLINICAL TRIAL: NCT03113409
Title: Buprenorphine as Adjunct to Outpatient Induction Onto Vivitrol
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: no funding available to continue
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Adam Bisaga, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #7456
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Opioid-use Disorder
Keywords: Outpatient detoxification; Opioid dependence; Naltrexone; Vivitrol; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Naltrexone; vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Procedure 1 (Experimental): Procedure 1: 5-day induction with increasing doses of oral naltrexone. Participants will receive XR-NTX on day five together with buprenorphine, and will continue receiving buprenorphine for 4 weeks until they receive 2nd XR-NTX dose.
  Interventions: Drug: Buprenorphine; Drug: Naltrexone; Drug: Vivitrol
- Procedure 2 (Experimental): Procedure 2: 10-day induction with buprenorphine administered daily and increasing daily doses of oral naltrexone beginning on day 2 . On day 10 participants will receive XR-NTX dose, and another one 4 weeks later. No buprenorphine will be given beyond day 10.
  Interventions: Drug: Buprenorphine; Drug: Naltrexone; Drug: Vivitrol
- Procedure 3 (Experimental): Procedure 3: 10-day induction with buprenorphine administered daily and increasing daily doses of oral naltrexone beginning on day 2 . On day 10 participants will receive XR-NTX dose, and another one 4 weeks later. Buprenorphine will continue for 4 weeks until the 2nd XR-NTX dose.
  Interventions: Drug: Buprenorphine; Drug: Naltrexone; Drug: Vivitrol

INTERVENTIONS:
Drug: Buprenorphine — Buprenorphine will be administered daily
Drug: Naltrexone — On study day 2, participants will receive increasing doses of oral naltrexone prior to administration of XR-NTX
Drug: Vivitrol — Participants will receive one 380 i.m. injection on Study day 5 or 10, and another injection 4 weeks later.
  Other Names: XR-NTX

SUMMARY:
The study will enroll 30 opioid-dependent participants into an open-label pilot outpatient study of methods to facilitate induction and stabilization onto XR-NTX. There will be three different methods of XR-NTX induction using increasing doses of oral naltrexone and buprenophine.

DETAILED DESCRIPTION:
Procedure 1: 5-day induction with increasing doses of oral naltrexone. Participants will receive XR-NTX on day five together with buprenorphine, and will continue receiving buprenorphine for 4 weeks until they receive 2nd XR-NTX dose.

Procedure 2: 10-day induction with buprenorphine administered daily and increasing daily doses of oral naltrexone beginning on day 2 . On day 10 participants will receive XR-NTX dose, and another one 4 weeks later. No buprenorphine will be given beyond day 10.

Procedure 3: 10-day induction with buprenorphine administered daily and increasing daily doses of oral naltrexone beginning on day 2 . On day 10 participants will receive XR-NTX dose, and another one 4 weeks later. Buprenorphine will continue for 4 weeks until the 2nd XR-NTX dose.

All participants will receive weekly therapy with a study psychiatrist. All participants will receive open-label medication.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60.
2. Meets DSM-5 criteria for current opioid use disorder (moderate-severe) of at least six months duration, supported by urine toxicology OR COWS score > or =6 OR Naloxone Challenge.
3. Voluntarily seeking treatment for opioid dependence.
4. In otherwise good health based on complete medical history and physical examination within normal ranges (AST or ALT < 3 times normal). )
5. Able to give written informed consent.

Exclusion Criteria:

1. Methadone maintenance treatment or regular use of illicit methadone (> 30 mg per week).
2. Maintenance on, or regular use of buprenorphine or other long-acting narcotic agonists.
3. Pregnancy, lactation, or failure in a sexually active woman to use adequate contraceptive methods.
4. Active medical illness which might make participation hazardous, such as untreated hypertension, acute hepatitis with AST or ALT > 3 times normal, AIDS (CD4 count under 200 currently or medically ill with an opportunistic infection), unstable diabetes.
5. Active psychiatric disorder which might interfere with participation or make participation hazardous, including DSM-5 Schizophrenia or any psychotic disorder, severe Major Depressive Disorder, or suicide risk or 1 or more suicide attempts within the past year.
6. Physiologically dependent on alcohol or sedative- hypnotics with impending withdrawal. Other substance use diagnoses are not exclusionary.
7. History of allergic or adverse reaction to buprenorphine, naltrexone, naloxone, clonidine, or clonazepam.
8. Chronic organic mental disorder (e.g. AIDS (CD4 count under 200 currently or medically ill with an opportunistic infection) dementia).
9. History of accidental drug overdose in the last 3 years as defined as an episode of opioid-induced unconsciousness or incapacitation, whether or not medical treatment was sought or received.
10. Painful medical condition that requires ongoing opioid analgesia or anticipated surgery necessitating opioid medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Procedure 1 | Procedure 2 | Procedure 3
Started | 10 | 0 (Study procedure was never started) | 0 (Study procedure was never started)
Completed | 5 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Procedure 1
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 34.5 [24 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 3
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Receive the Second Injection of XR-NTX.
Description: Percentage of patient who initiated Procedure 1 and completed the study receiving the 2nd injection of XR-NTX
Time Frame: 4 weeks after 1st injection
Population: all participants enrolled in the study (Procedure 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Procedure 1
Number analyzed (Participants) | 10
Participants | 6

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: AE data were collected over the period of study participation, which is 8 weeks for each participant
Arm/Group | Procedure 1
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT03113409/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT03113409/SAP_001.pdf